CLINICAL TRIAL: NCT02107690
Title: The Influence of Lidocaine Temperature on Pain During Subcutaneous Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/2297
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Needlestick Injuries
Keywords: Injections; Temperature; Pain; Healthy volunteers; Lidocaine
MeSH Terms: conditions — Needlestick Injuries; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- low temperature (Experimental): Each participant will receive three lidocaine injections subcutaneously on the abdomen at different temperatures
  Interventions: Procedure: Low temperature lidocaine injection
- room temperature (Experimental): Each participant will receive three lidocaine injections subcutaneously on the abdomen at different temperatures
  Interventions: Procedure: Room temperature lidocaine injection
- body temperature (Experimental): Each participant will receive three lidocaine injections subcutaneously on the abdomen at different temperatures
  Interventions: Procedure: Body temperature lidocaine injection

INTERVENTIONS:
Procedure: Low temperature lidocaine injection — 4 °C
  Arms: low temperature
Procedure: Room temperature lidocaine injection — 20 °C
  Arms: room temperature
Procedure: Body temperature lidocaine injection — 37 °C
  Arms: body temperature

SUMMARY:
This study will investigate the influence of lidocaine temperature on pain during injection of lidocaine. Each participant will receive three injections subcutaneously on the abdomen with different temperatures. After each injection, participants will be asked to evaluate the pain on a Visual analog scale (0-100 mm). It is anticipated that the pain decreases with increasing temperature. The aim of the study is to find a simple method for pain reduction that can be used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years

Exclusion Criteria:

* Kidney, heart or liver disease
* Eczema or psoriasis on injection site
* Neuropathy
* Regular use of painkillers
* Hypersensitivity of Lidocaine
* Pregnancy
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pain | 60 seconds
  (1) visual analog scale 0-100mm, (2) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, prof md, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lundbom JS, Tangen LF, Wago KJ, Skarsvag TI, Ballo S, Hjelseng T, Foss OA, Finsen V. The influence of Lidocaine temperature on pain during subcutaneous injection. J Plast Surg Hand Surg. 2017 Apr;51(2):118-121. doi: 10.1080/2000656X.2016.1194281. Epub 2016 Jun 17. PMID 27314148